CLINICAL TRIAL: NCT07004634
Title: Comparison of the Application Effects of Different Drainage Modes in the Perioperative Period of Minimally Invasive Three-Field Radical Esophagectomy for Esophageal Cancer
Brief Title: Comparison of Drainage Methods in Minimally Invasive Esophagectomy (DEMURE）
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RTS-026
Record Dates: First submitted 2025-05-05; First posted 2025-06-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Cancer; Drainage/Methods; Postoperative Pain
Keywords: Esophageal cancer; Mediastinal drainage tube; Postoperative pain
MeSH Terms: conditions — Esophageal Neoplasms; Pain, Postoperative | interventions — Chest Tubes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abdominal mediastinal tube (Experimental): Transperitoneal mediastinal drainage was performed for postoperative management of the patient.
  Interventions: Procedure: Abdominal mediastinal tube
- Chest mediastinal tube (Experimental): Transthoracic mediastinal drainage was performed for postoperative management of the patient.
  Interventions: Procedure: Chest mediastinal tube
- Chest tube + chest mediastinal tube (Experimental): Chest tube insertion combined with transthoracic mediastinal drainage was performed for postoperative management of the patient.
  Interventions: Procedure: Chest tube + chest mediastinal tube

INTERVENTIONS:
Procedure: Chest mediastinal tube — Transthoracic mediastinal drainage was performed for postoperative management of the patient.
  Arms: Chest mediastinal tube
Procedure: Abdominal mediastinal tube — Transperitoneal mediastinal drainage was performed for postoperative management of the patient.
  Arms: Abdominal mediastinal tube
Procedure: Chest tube + chest mediastinal tube — Chest tube insertion combined with transthoracic mediastinal drainage was performed for postoperative management of the patient.
  Arms: Chest tube + chest mediastinal tube

SUMMARY:
This RCT compares three drainage approaches after minimally invasive esophagectomy (chest tube + thoracic mediastinal drainage tube, thoracic, and abdominal mediastinal drainage tube) to evaluate perioperative outcomes, addressing current evidence gaps in pain and complication profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Pathologically confirmed esophageal cancer requiring three-incision esophagectomy (cervical, thoracic, and abdominal incisions)
* ASA physical status class I-III

Exclusion Criteria:

* History of chronic pain or long-term use of analgesics prior to surgery
* Severe cardiopulmonary dysfunction (e.g., FEV1 <50%)
* Coagulation disorders or patients undergoing reoperation
* Intraoperative findings of extensive pleural adhesions, combined resection of adjacent organs, or other conditions deemed by the investigator to warrant exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Scores | Pain scores were recorded at different times during the postoperative period when the patients were quiet and active (at 7 AM, 11 AM, 3 PM, and 7 PM) from postoperative day 1 to postoperative day 4.
  Pain scores were assessed based on the visual analog scale according to the World Health Organization guidelines, in which 0 indicated no pain and 10 indicated the worst possible pain.
  We also recorded and evaluated maximum daily pain scores when pain caused by the mediastinal drainage tube incision.

SECONDARY OUTCOMES:
Postoperative complications | Postoperative complications from posoperative day 1 to postoperative month 3
  Postoperative complications included anastomotic leak, major pulmonary complications, and major abdominal complications. Pleural effusion was defined as a drainage volume of greater than 800 mL. Pneumothorax was defined by a distance of greater than 3 cm between the apex of the lung and the top of the ribcage on chest radiography.

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, PhD, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified baseline characteristics, outcomes, and adverse events.